CLINICAL TRIAL: NCT00889135
Title: Long Term Treatment With L-DOPS
Status: Approved for marketing | Type: Expanded Access
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, David Robertson, Professor of Medicine and Pharmacology, Vanderbilt University
Other Study IDs: 041037
Record Dates: First submitted 2009-04-24; First posted 2009-04-28 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Dopamine Beta Hydroxylase (DBH) Deficiency
MeSH Terms: interventions — Droxidopa

INTERVENTIONS:
Drug: droxidopa — Droxidopa (L-DOPS) comes in capsule form, 100 mg or 200 mg strength and is usually administered 2 - 3 times per day. It would be taken indefinitely to improve symptoms of orthostatic hypotension
  Other Names: L-DOPS; DOPS

SUMMARY:
This study is designed to supply L-DOPS (droxidopa) on a long term basis to patients with a genetic form of profound orthostatic hypotension, most commonly DBH deficiency. It also allows us to collect medical history information on this small population of patients that would allow us to determine if there are any complications from this type of treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older with orthostatic hypotension
* established diagnosis of DBH deficiency and fractionated plasma catecholamine levels that show high dopamine levels and very low norepinephrine and epinephrine levels. Blood pressure increase in response to oral treatment with L-DOPS during previous studies.

Exclusion Criteria:

* subjects with orthostatic hypotension that do not have a genetic form of the disorder and catecholamine pattern is not consistent with that above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Robertson, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States